CLINICAL TRIAL: NCT06837896
Title: A Multicenter Study Evaluating the Efficacy and Safety of QLG1080 in Patients With Hormone-sensitive Advanced Prostate Cancer
Brief Title: Efficacy and Safety Study of QLG1080 in Patients With Hormone-sensitive Advanced Prostate Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLG1080-301
Record Dates: First submitted 2025-02-17; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLG1080 (Experimental)
  Interventions: Drug: QLG1080

INTERVENTIONS:
Drug: QLG1080 — Oral administration

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of QLG1080 in patients with hormone-sensitive advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histological or cytological diagnosis of prostate cancer;；
* Advanced prostate cancer patients eligible for endocrine therapy, able to receive continuous androgen deprivation therapy for at least 6 months.
* Serum testosterone ≥150 ng/dL (5.2nmol/L) at screening visit;
* The Eastern Cooperative Oncology Group (ECOG) score is 0 to 1.

Exclusion Criteria:

* Diagnosed or suspected of hormone-resistant prostate cancer;
* For prostate cancer patients who have had or are undergoing endocrine therapy
* Patients who have previously undergone pituitectomy or adrenalectomy or have pituitary disease or adrenal dysfunction;
* Those who have had any prostate surgery within 4 weeks prior to initial dosing or prostate surgery or other major surgical treatment during the planned trial period (except urinary tract obstruction relief);
* The imaging results of screening visits clearly showed the presence of brain metastases;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sustained castration rate of serum testosterone | From study day 29 to the end of the study
  The cumulative probability of serum testosterone levels reaching and maintaining castration levels (≤50 ng/dL or 1.7 nmol/L)